CLINICAL TRIAL: NCT00627289
Title: The Effect of Selective Neurectomy and Mesh Removal on Chronic Postherniotomy Pain
Brief Title: Selective Neurectomy and Mesh Removal for Chronic Postherniotomy Pain
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, M.D., Rigshospitalet, Denmark
Other Study IDs: (KF) 11 320499.
Record Dates: First submitted 2008-02-12; First posted 2008-03-03 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2012-10

CONDITIONS: Pain
Keywords: Chronic pain; groin hernia; neuropathic pain; chronic postoperative pain; Postherniotomy pain; Neuroplastic changes
MeSH Terms: conditions — Pain; Chronic Pain; Hernia, Inguinal; Neuralgia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients with chronic postherniotomy pain (>1 year), affecting everyday activities severely

SUMMARY:
Chronic postherniotomy pain affects every day activities in 5-8% of patients. However, no established treatment for this pain syndrome exists and previous reports on the effect of surgical intervention suffer from methodological problems. The neurophysiological characteristics suggest that pain arises from deeper neuronal structures injured during surgery or by ongoing inflammation from the mesh. This study investigates the effect of removing inserted mesh and compressed nerves on pain related daily impairment of activities assessed by the validated AAS questionnaire before and 6 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult ( more than 18 years old) patients with chronic pain after groin hernia surgery, and pain related impairment of everyday function. The pain should have occurred after previous open surgery.
* The patient should be able to locate to a specific area with maximum pain. Patients should be able to understand and use pain scales, and the AAS-scale.

Exclusion Criteria:

* All that contradicts the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain occuring after groin hernia repair. Patients must experience moderate/severe pain related impairment of everyday activities. Patients have to be able to localize a maximum point of pain.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
changes in AAS scores before and six months after operation | 6 months

SECONDARY OUTCOMES:
changes in sensory function assessed by quantitative sensory testing | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, M.D., Study Director — Rigshospitalet, Copenhagen University, Denmark; Henrik Kehlet, M.D., Ph. D., Principal Investigator — Rigshospitalet, Copenhagen University, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Ambulatory Surgical Clinic, Hørsholm Hospital, Hørsholm

REFERENCES:
- [Background] Aasvang E, Kehlet H. Surgical management of chronic pain after inguinal hernia repair. Br J Surg. 2005 Jul;92(7):795-801. doi: 10.1002/bjs.5103. PMID 15962258